CLINICAL TRIAL: NCT03138408
Title: An Open Label, Phase 1 Study of SC-004 as Monotherapy and in Combination With ABBV-181 in Subjects With Epithelial Ovarian, Including Fallopian Tube and Primary Peritoneal and Endometrial Cancers
Brief Title: SC-004 Alone or With ABBV-181 in Subjects With Epithelial Ovarian, Fallopian Tube, Primary Peritoneal and Endometrial Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M16-553
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Cancer
Keywords: Ovarian cancer; Endometrial cancer; SC-004; Maximum tolerated dose (MTD); ABBV-181
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms | interventions — SC004; budigalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SC-004 (Experimental)
  Interventions: Drug: SC-004
- SC-004 and ABBV-181 (Experimental)
  Interventions: Drug: SC-004; Drug: ABBV-181

INTERVENTIONS:
Drug: SC-004 — Intravenous
Drug: ABBV-181 — Intravenous
  Arms: SC-004 and ABBV-181

SUMMARY:
This is a two-part study consisting of Part A (dose regimen finding) followed by Part B (dose expansion). Part A (dose regimen finding) will allow definition of the maximum tolerated dose (MTD) through dose escalation and possible dose interval modification. In Part B (dose expansion), potential therapeutic doses may be studied with SC-004 as monotherapy and SC-004 in combination with ABBV-181 in disease-specific cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced malignancy defined as any of the following tumors for which no further standard or curative therapy exists or is considered appropriate by the Investigator:

  * Epithelial ovarian cancer, including fallopian tube cancer or primary peritoneal cancer, of high-grade serous histology, with platinum refractory or resistant disease after prior treatment with at least one platinum-based chemotherapeutic regimen. In Part B (dose expansion), subjects may have received no more than 3 lines of systemic cytotoxic chemotherapy.

    * Note, the line of therapy limit does not apply to the biopsy substudy cohorts.
  * Metastatic or advanced endometrial carcinoma previously treated with at least 1 platinum-based chemotherapeutic regimen.
* Eastern Cooperative Oncology Group (ECOG) 0-1.
* Adequate hematologic, hepatic, and renal function.

Exclusion Criteria:

* Participants with prior exposure to a pyrrolobenzodiazepine or indolinobenzodiazepine based drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities (DLT) | Minimum first cycle of dosing (21-day cycles)
  DLTs graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.

SECONDARY OUTCOMES:
Observed plasma concentrations at trough (Ctrough) | Approximately 1 year
  Observed plasma concentrations at trough.
Overall Survival (OS) | Approximately 2 years
  OS is defined as the time from the subject's first dose date to death due to any cause.
Objective Response Rate (ORR) | Approximately 2 years
  ORR is defined as the proportion of subjects with complete response or partial response (CR+PR).
Terminal half life (T1/2) | Approximately 1 year
  Terminal half life (T1/2).
Maximum observed serum concentration (Cmax) | Approximately 1 year
  Maximum observed serum concentration.
Time to Cmax (Tmax) | Approximately 1 year
  Time to Cmax.
Clinical Benefit Rate (CBR) | Approximately 2 years
  CBR is defined as the proportion of subjects with an objective response or stable disease (CR+PR+SD).
Progression Free Survival (PFS) | Approximately 2 years
  PFS time is defined as the time from the subject's first dose of study drug (Day 1) to either the subject's disease progression or death due to any cause, whichever occurs first. Under the situation that neither event occurs, the PFS time will be censored at the date of last tumor assessment. Subjects lacking an evaluation of tumor response after their first dose of study treatment will have their event time censored at Day 1.
Duration of Response (DOR) | Approximately 2 years
  DOR is defined as the time from the subject's initial objective response (CR or PR) to study drug therapy to disease progression or death due to any cause, whichever occurs first. If the dates of disease progression or death are not available, the DOR will be censored at the date of last valid tumor assessment.
Area under the plasma concentration-time curve within a dosing interval (AUC) | Approximately 1 year
  Area under the plasma concentration-time curve within a dosing interval.
QTcF Change from Baseline | Up to 9 weeks based on 3 cycles of dosing (21-day cycles)
  QT interval measurement corrected by Fridericia's formula (QTcF).
Duration of Clinical Benefit (DOCB) | Approximately 2 years
  DOCB is defined as the time from a subject's objective response (CR or PR) or stable disease (SD) to study drug therapy to disease progression or death due to any cause whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (12):
- United States (12):
  - University of Alabama /ID# 202249, Birmingham, Alabama
  - Highlands Oncology Group /ID# 209165, Fayetteville, Arkansas
  - City of Hope /ID# 202493, Duarte, California
  - University of Chicago /ID# 200735, Chicago, Illinois
  - Henry Ford Health System /ID# 202480, Detroit, Michigan
  - Mayo Clinic - Rochester /ID# 200732, Rochester, Minnesota
  - Washington University School /ID# 164091, St Louis, Missouri
  - The Ohio State University - Columbus /ID# 164089, Columbus, Ohio
  - Univ Oklahoma HSC /ID# 164090, Oklahoma City, Oklahoma
  - Tennessee Oncology-Nashville Centennial /ID# 164088, Nashville, Tennessee
  - MD Anderson Cancer Center /ID# 200048, Houston, Texas
  - Huntsman Cancer Institute /ID# 209164, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No